CLINICAL TRIAL: NCT00721019
Title: Sleep, Energy Metabolism and Diabetes Risk.
Brief Title: Sleep Loss and Glucose Metabolism in People With Family History of Type 2 Diabetes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 16079A-S3; R01HL089637 (NIH)
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Sleep; Sleep Deprivation; Insulin Resistance; Type 2 Diabetes
Keywords: short sleep duration; glucose clamp technique; insulin secretion; insulin action; lipid turnover; free fatty acids
MeSH Terms: conditions — Sleep Deprivation; Insulin Resistance; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5-hour bedtime (Experimental)
  Interventions: Other: 5-hour bedtime
- 8.5-hour bedtime (Experimental)
  Interventions: Other: 8.5-hour bedtimes

INTERVENTIONS:
Other: 5-hour bedtime — 10 days with sleep restricted only to a 5-hour bedtime period at night
  Arms: 5-hour bedtime
Other: 8.5-hour bedtimes — 10 days with sleep allowed only during a 8.5-hour period at night
  Arms: 8.5-hour bedtime

SUMMARY:
The use of sugar and starch-like foods for energy (carbohydrate metabolism) changes when people sleep. However, it is still not known if differences in the amount of nighttime sleep have an effect on the carbohydrate metabolism of people who have a relative with type 2 diabetes (parent, sibling, or grandparent). This study is being done to test the hypothesis that the carbohydrate metabolism of people who have a history of type 2 diabetes in their family will be different after they have slept short hours for 10 days in comparison to when they have slept longer hours for 10 days.

DETAILED DESCRIPTION:
Study participants will complete two 10-day inpatient stays in the sleep laboratory of the University of Chicago Clinical Resource Center scheduled at least 4 weeks apart. Bedtime duration will be set at 5 hours per night during one of these stays and 8.5 hours per night during the other. No daytime naps will be allowed. Study participants will be served regular daily meals including breakfast, lunch, dinner, and a bedtime snack. On weekdays all participants will engage in simulated "office work" while in the sleep laboratory. During the rest of the time participants will maintain their usual indoor and outdoor activities as much as possible within the limits of the University of Chicago campus. During the last two days of each inpatient stay in the laboratory, participants will undergo two different tests. The first test will determine how much insulin does their body produce in response to an intravenous glucose infusion lasting several hours. The second test will determine how effective is the action of the sugar-processing hormone, insulin, in their body when it is infused intravenously together with glucose over a period of several hours.

ELIGIBILITY:
Inclusion Criteria:

* regular sleep habits
* BMI 20 to 27 kg/m2
* at least one parent, sibling or grandparent with type 2 diabetes
* no regular exercise habits

Exclusion Criteria:

* active smoker
* night or shift work
* have highly variable sleep habits
* have a hormonal disorder
* have a sleep disorder
* have an active medical problem
* women only: use of birth control pills
* women only: irregular menstrual periods or pregnancy
* use of medications/compounds that can disrupt sleep

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2008-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Total body insulin sensitivity | at the end of each bedtime intervention

SECONDARY OUTCOMES:
First and second phase insulin secretion | at the end of each bedtime intervention
Endogenous glucose production | at the end of each bedtime intervention
Glycerol turnover and free fatty acid concentrations | at the end of each bedtime intervention

CONTACTS AND LOCATIONS:
Overall Officials: Plamen D Penev, MD, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States